CLINICAL TRIAL: NCT01533129
Title: Phase 4 Study That Evaluates the Effects of Two Different Testosterone Replacement Regiments on Endothelial Dysfunction, Inflammation and Insulin Resistance in Male Subjects With Hypogonadotrophic Hypogonadism.
Brief Title: The Effect of Testosterone Replacement on Endothelial Dysfunction, Inflammation and Insulin Resistance in Male Hypogonadotrophic Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Alper Sonmez, Associate Professor in Medicine, Gulhane School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSM-022011
Record Dates: First submitted 2011-12-13; First posted 2012-02-15 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Hypogonadotrophic Hypogonadism
Keywords: Hypogonadism; Endothelial dysfunction; Inflammation; Insulin resistance; Testosterone replacement therapy
MeSH Terms: conditions — Hypogonadism; Inflammation; Insulin Resistance | interventions — Testosterone; Injections; Adenosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily testosterone transdermal gel (Active Comparator)
  Interventions: Drug: Testogel 50 mg transdermal gel
- Injectable Testosterone esters (Active Comparator): Testosteron 250mg injection per 3-4 weeks for 6 months
  Interventions: Drug: Testosterone 250mg injection

INTERVENTIONS:
Drug: Testogel 50 mg transdermal gel — 50mg testosterone gel implementation on every night
  Other Names: Testogel 50mg transdermal gel
  Arms: Daily testosterone transdermal gel
Drug: Testosterone 250mg injection — The testosterone 250mg ester IM injections performed in three weeks.
  Other Names: Sustanon 250 mg amp.
  Arms: Injectable Testosterone esters

SUMMARY:
The study searched for answers to two questions

1. What is the effect of testosterone replacement therapy on endothelial dysfunction, inflammation and insulin resistance?
2. Regarding the above parameters, is there any difference between daily transdermal testosterone implementation and intramuscular injection performed in three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Treatment naive
* Hypogonadotrophic hypogonadism

Exclusion Criteria:

* Previous history of androgen replacement
* Chronic metabolic disorders

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The alterations in the measures for endothelial functions | 6 months
  The alterations in Endothelial functions are determined by measuring plazma ADMA levels, as a surrogate. ADMA measurement is pereformed by ELISA kit (Immundiagnotik, Bensheim, Germany)(Catalog Number 7828) with a minimal detection limit of 0.05µmol/L.
The alterations in the measures of insulin resistance | 6 months
  The alterations in insulin sensitivity are estimated by using the HOMA index by the formula, HOMA-IR = (insulin x glucose)/405.
The alterations in the measures of inflammation | 6 months
  The alterations in the measures of inflammation are determined by measuring Human Pentraxin-3 levels. ELISA kiti /R&D Systems, Inc. Minneapolis, MN, ABD) (Catalog number DPTX30) with a minimal detection limit of 0.025ng/ml, intraassay CV of 3.8-4.4%, and interassay CV of 4.1-6.1% was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine Department of Endocrinology and Metabolism, Ankara, Non US, Turkey (Türkiye)